CLINICAL TRIAL: NCT03852381
Title: Mechanisms and Outcome-Prognostication for Paresthesia-based and -Free Spinal Cord Stimulation in Patients With Persistent Neuropathic Pain: the MOPPStim Study
Brief Title: Mechanisms and Outcome-Prognostication for Paresthesia-based and -Free Spinal Cord Stimulation
Acronym: MOPPStim
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: MSH-UHN AMO Innovation Fund (Unknown)
Responsible Party: Principal Investigator, Anuj Bhatia, Director, Anesthesia Chronic Pain Clinical Services, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-5864
Record Dates: First submitted 2018-12-31; First posted 2019-02-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Neuropathic Pain; Chronic Pain
Keywords: Spinal Cord Stimulation; Burst Stimulation; High Frequency Stimulation; High Density Stimulation; fMRI; MEG; QST
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Spinal Cord Stimulation (Experimental): At baseline, the following data will be recorded: standard-of-care questionnaire scores, neuroimaging (fMRI, MEG), psychophysical testing (QST), accelerometer sleep and activity data.
  The trial will proceed as follows:
  Day 1-4: Paresthesia-based SCS (PB-SCS)
  Day 5-8: No SCS (placebo)
  Day 9-12: PF-SCS
  Neuroimaging and psychophysical testing will be conducted at the end of the trial, and will be assessed 6-months post-implantation of the SCS device along with adverse effects. A decision to implant the SCS system will be made based on reduction of patient pain intensity by 50% in PB-SCS and/or PF-SCS modes, but not with placebo SCS.
  Based on the response in the trial, the patient will either not be a candidate for an SCS implant, or they will receive one of the four modes upon implantation (PB-SCS, or one of the three PF-SCS: Burst, High Frequency, High Density).
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Paresthesia-based SCS(PB-SCS), with stimulating frequencies between 30 to 80 Hz that confer a tingling sensation. Three different paresthesia-free SCS (PF-SCS) modes that use frequencies in the range of 400-10,000 Hz include Burst, High Frequency stimulation at 1.2 kHz and High Density stimulation at 400 Hz.

SUMMARY:
Spinal cord stimulation (SCS) relies on stimulation of pain-relieving pathways in the spinal cord to treat chronic neuropathic pain. Traditional paresthesia-based SCS (PB-SCS) relies on providing analgesia through stimulation of spinal cord dorsal columns but it is often associated with attenuation of analgesic benefit and lack of acceptance of paresthesias. Recently introduced three different paresthesia-free (PF-SCS) modes of stimulation aim to overcome limitations of PB-SCS. Several questions regarding PB and PF SCS modes remain unanswered including the mechanisms of therapeutic benefit, criteria for selecting patients likely to benefit, and long-term outcomes. A concerted effort is required to understand and optimize utilization of SCS. This project has the twin goals of using neuroimaging techniques to understand mechanisms that underlies analgesic benefit from PB/PF-SCS modes and to identify criteria for selecting patients based on monitoring of pain and its related domains in patients undergoing SCS trials. Achieving these objectives will increase probability of analgesic benefit while minimizing adverse effects and knowledge gains from this study will be applicable to other therapies for chronic pain conditions.

DETAILED DESCRIPTION:
Over 7 million Canadians suffer from chronic pain with 1 in 4 patients having neuropathic pain (NP), a condition caused by injury to nerves in the body. NP tends to have an extremely unpleasant character, severe intensity, and a persistent unremitting course. Conventional medical management (CMM) is often ineffective in relieving NP in majority of these patients. Paresthesia-Based Spinal Cord Stimulation (PB-SCS) has been used to treat NP but it has limitations in terms of preserving analgesic benefit and it is often associated with adverse effects. Recently introduced Paresthesia-Free SCS (PF-SCS), available at all tertiary level pain centers, has the potential to overcome these limitations but knowledge gaps remain in understanding and applying this modality.

The study design will be a prospective, exploratory study with randomization of order of no stimulation with novel modes of PF-SCS during the SCS trial and blinding of subjects (as per clinical standard of care) and outcome assessors. Participants with appropriate indications for trial of SCS with novel paresthesia-free modes will be enrolled. Baseline demographic and pain-related data including opioid intake in Oral Morphine Equivalents Per day in mg (OMED) will be collected. Pre-SCS trial neuroimaging (fMRI, MEG) and QST will be performed to establish parameters for future comparisons. Data on physical activity and sleep will be collected using actigraphy, as per standard of care. Data on pain and its related domains will be collected using validated questionnaires on the Manage My Pain app, in which all questionnaires administered are part of the patient's clinical standard of care. Ninety subjects will undergo a percutaneous trial of SCS that will last 12 days and the trial will be divided into three phases. All subjects will trial a conventional paresthesia-based SCS mode in the first four days of the trial. Subjects will then proceed the next four days (day 5-8) with no (placebo) stimulation, followed by one of the three novel PF-SCS modes (Burst, High Frequency, High Density) for the last 4 days of the trial. This process is currently adopted for all patients receiving SCS as standard of care. Neuroimaging (fMRI, MEG) and QST will be performed at the end of the SCS trial. Subjects who achieve significant reduction in pain, disability and sleep disturbance questionnaire scores with one of the novel PF-SCS modes will be offered percutaneous implantation of SCS system 4 to 6 weeks after the end of the trial using the novel PF-SCS mode they experienced during the trial. MEG and QST will be performed and data from validated questionnaires on the Manage My Pain app will be collected at 6 months after implantation.

Use of fMRI (functional Magnetic Resonance Imaging), MEG (Magnetoencephalography), and QST (Quantitative Sensory Testing) in this study will help improve understanding of the alteration in brain in NP and the analgesic action of PB/PF-SCS. Validation of wearable technology and of app-based digital platforms will allow these available but infrequently-used modalities to improve success of analgesic treatments in patients with chronic pain. Healthcare systems will benefit through efficient use of resources to treat chronic pain made possible by understanding what works, who does it work for, and how to predict analgesic benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 - 80 years of age, with refractory neuropathic pain (as per clinical features and DN4 score > 3/10) in back and or lower limbs for more than 3 months following lumbar spine surgery
2. Severity of pain > 3/10 on NRS and ODI score for disability >40/100; and
3. Pain refractory to conventional medical management tried for at least 3 months.

Exclusion Criteria:

1. Age < 18 or age ≥ 80 years;
2. Previous trial or implantation of SCS system;
3. Procedural contraindications to SCS including extensive thoracolumbar spine surgery, moderate-to-severe central canal stenosis, coagulopathy, local or systemic infection;
4. Pregnancy;
5. Opioid dose > 200 mg OMED;
6. Psychiatric or psychological disorder likely to impact perception of pain;
7. Inability to comply with the study interventions or evaluate treatment outcomes;
8. Mechanical spine instability as per flexion/extension lumbar X-rays;
9. Ongoing litigation issues related to the pain; and
10. Concomitant peripheral neuropathy or myopathy or central neuropathic pain (e.g. post-stroke pain).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in neuronal activity with the novel PF-SCS modes as detected by fMRI and MEG | 12 days after the initiation of the SCS trials )
Changes in neuronal activity with the novel PF-SCS modes as detected by fMRI and MEG | 6 months after the initiation of the SCS implants
To measure long-term outcomes of novel PF-SCS modes including intensity and quality of pain, physical and psychological functioning, and patients' global impression of change | 6 months after the initiation of the SCS implants.
Changes in sensory threshold with the novel PF-SCS modes as detected by QST | 6 months after the initiation of the SCS implants

SECONDARY OUTCOMES:
To measure incidence of more than 50% reduction in pain intensity scores in patients with NP syndromes with novel modes of SCS | Six months after implantation.
To correlate data on physical activity as measured by an accelerometer during trials of novel SCS modes with data obtained from validated questionnaires | 12 days after the initiation of the SCS trial
To correlate data on sleep as measured by an accelerometer during trials of novel SCS modes with data obtained from validated questionnaires | 12 days after the initiation of the SCS trial
To measure incidences of analgesic failure (as indicated with less than 50% reduction in pain intensity scores) and adverse effects of PF-SCS | Six months after implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Feigin G, Dana E, Bains V, Bhatia A. Evaluating patient satisfaction and perceived accuracy in questionnaires completed before vs. during a pain clinic visit. Pain Manag. 2025 Sep;15(9):571-576. doi: 10.1080/17581869.2025.2529773. Epub 2025 Jul 7. PMID 40623913